CLINICAL TRIAL: NCT00052312
Title: Randomized Trial Of Adriamycin (A) Cisplatin (P) Chemotherapy Versus Paclitaxel (T) Adriamycin (A) And Cisplatin (P) In Patients With Metastatic/Relapsed Or Locally Advanced Inoperable Endometrial Cancer
Brief Title: Doxorubicin and Cisplatin With or Without Paclitaxel in Treating Patients With Locally Advanced, Metastatic, and/or Relapsed Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-55984; EORTC-55984
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; endometrial papillary serous carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cisplatin; Doxorubicin; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether doxorubicin and cisplatin are more effective with or without paclitaxel in treating endometrial cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of combining doxorubicin and cisplatin with or without paclitaxel in treating patients who have locally advanced, metastatic, and/or relapsed endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with locally advanced, metastatic, and/or relapsed endometrial cancer treated with doxorubicin and cisplatin with or without paclitaxel.
* Compare the toxicity of these regimens in these patients.
* Compare the progression-free survival at 18 months of patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to performance status (0 vs 1 vs 2), metastatic disease (M0 vs M1), prior pelvic radiotherapy for pelvic recurrence (yes vs no), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxorubicin IV over 30 minutes, paclitaxel IV over 3 hours, and cisplatin IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive doxorubicin and cisplatin as in arm I. Quality of life is assessed at baseline, before each course, after courses 3 and 6, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter. In the event of progressive disease, quality of life is assessed every 3 months.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter. In the event of progressive disease, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 140 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed endometrial epithelial carcinoma meeting at least 1 of the following criteria:

  * Advanced metastatic and/or relapsed disease
  * Locally advanced inoperable or unresectable disease
* No mixed mesodermal tumor and/or tumors showing evidence of sarcomatous elements
* Uterine papillary serous carcinoma allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL (transfusions allowed)

Hepatic

* ALT and AST less than 2 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2 times ULN
* Bilirubin less than 1.5 times ULN

Renal

* Creatinine less than 1.5 times ULN
* Creatinine clearance greater than 50 mL/min

Cardiovascular

* Normal baseline EKG
* Normal baseline LVEF on MUGA or echocardiogram for patients who received prior anthracyclines

Other

* Able to tolerate high-dose dexamethasone
* Must be considered fit for chemotherapy
* No uncontrolled infection
* No other malignancy within the past 5 years except successfully treated basal cell skin cancer or carcinoma in situ of the cervix
* No prior nervous or psychiatric disorder that would preclude study compliance
* No psychological, familial, sociological, or geographic condition that would preclude study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 12 months since prior adjuvant chemotherapy
* Total dose of prior doxorubicin no greater than 200 mg/m^2
* Total dose of prior epirubicin no greater than 300 mg/m^2

Endocrine therapy

* At least 28 days since prior hormonal therapy for patients with partial or complete response after first-line treatment

Radiotherapy

* No prior radiotherapy to any area other than pelvis
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent anticancer medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2002-09; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival as measured by Kaplan Meier and RECIST at 18 months

SECONDARY OUTCOMES:
Overall survival as measured by Kaplan Meier after each course, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter
Toxicity as measured by NCIC Common Toxicity Criteria v2.0 after each course

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S. Reed, MD, Study Chair — University of Glasgow; Giorgio Bolis, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (35):
- Allgemeines Krankenhaus - Universitatskliniken, Vienna, Austria
- Belgium (6):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - U.Z. Gasthuisberg, Leuven
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- France (2):
  - Centre Regional Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - Azienda Sanitaria Ospedaliera Ordine Mauriziano, Turin
  - Clinica Universitaria, Turin
  - Ospedale Civile, Voghera
- Netherlands (6):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Utrecht, Utrecht
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- Spain (3):
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto Valenciano De Oncologia, Valencia
- United Kingdom (11):
  - Royal United Hospital, Bath, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oldchurch Hospital, Romford, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - Western Infirmary, Glasgow, Scotland